CLINICAL TRIAL: NCT00867438
Title: Efficacy and Tolerability of a New Oral Extended-Release Formulation Containing Parnaparin Sodium (CB-01-05-MMX™), Administered as Add-on Therapy to Oral Mesalazine or Other 5-ASA Derivatives, in Patients With Active, Left-Sided, Mild to Moderate Ulcerative Colitis. A Multicentre Randomized, Double-Blind, Comparative Study Versus Placebo.
Brief Title: Efficacy and Tolerability of a New Oral Extended-Release Formulation Containing Parnaparin Sodium, Administered Add-on Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cosmo Technologies Ltd (Industry)
Responsible Party: Cosmo Technologies Ltd, Cosmo Technologies Ltd
Organization: CosmoTech (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CB-01-05/04
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis; Left-sided, mild to moderate ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Sigmoidoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Procedure: Sigmoidoscopy
- 2 (Experimental)
  Interventions: Procedure: Sigmoidoscopy

INTERVENTIONS:
Procedure: Sigmoidoscopy

SUMMARY:
The objective of this study is to evaluate the efficacy and the tolerability of oral parnaparin sodium (210mg), administered in extended-release tablets identified as CB-01-05-MMX™.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients, between 18 and 70 years of age.
2. Patients with a confirmed diagnosis of ulcerative colitis in treatment with fixed-dose of oral mesalazine or other 5-ASA derivatives for at least 4 weeks with a high clinical suspicion of active disease, confirmed by sigmoidoscopy at enrolment in the study .
3. Presence of ulcerative colitis located at left side of the colon, from splenic flexure of the colon to the rectum (up to 15 cm proximal to the anus).
4. Patients with mild to moderate active ulcerative colitis, as defined by the DAI ≥ 4 and ≤ 10, and CAI ≥ 5 and ≤ 12.
5. Women with negative serum test for pregnancy.
6. Women of childbearing potential provided they use adequate contraceptive precautions during the treatment period. Adequate contraceptive methods are defined as those with a failure rate <1% per year when correctly used, and include implants, injectables, combined oral pills, some IUDs or a vasectomised partner in a stable relationship.
7. Ability to understand and willing to sign the Informed Consent Form, and other documents required to be read or signed by the subject.

Exclusion Criteria:

1. Presence of other clinically significant medical condition as determined by the Investigator.
2. History of hypersensitivity or idiosyncratic reaction to heparins.
3. History of hemorrhages, excluding intestinal bleeding due to ulcerative colitis, hemocoagulative disorders, or platelet dysfunction.
4. Presence of arterial hypertension (SAP ≥ 160 mm Hg; DAP ≥ 95 mm Hg).
5. Receipt of any investigational agent within 90 days of starting treatment.
6. Use of rectal 5-ASAs or rectal corticosteroids within 2 weeks before the starting the study.
7. Use of anti-TNF agents or immunosuppressive drugs such as azothioprine, 6-mercaptopurine or cyclosporine A in the last 3 months.
8. Patients with ulcerative colitis of severe entity (DAI > 10 or CAI > 12), or with limited distal ulcerative proctitis, or with infectious colitis confirmed by microbiological assessment in stool.
9. Patients with severe intestinal bleeding, or with Hb < 9 g/dL.
10. Presence of significant hepatic impairment (AST, ALT > 2 ULN).
11. Presence of significant renal impairment (creatinine > 2 ULN).
12. Women who are pregnant or who are breast feeding.
13. Intestinal obstruction.
14. Presence of type 1 or type 2 diabetes.
15. Concomitant oral antibiotic treatment, within 2 weeks before starting the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The number of patients achieving clinical remission (CAI <4). | 8 weeks

SECONDARY OUTCOMES:
Endoscopic Index, Histologic Score of mucosal bioptic specimens, AEs, laboratory parameters, vital signs. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gasbarrini, Prof, Principal Investigator — Department of Internal Medicine